CLINICAL TRIAL: NCT04943965
Title: Repeatability, Reproducibility, and Efficacy Testing of Automated Hemodynamic Output by Transthoracic Echocardiography
Brief Title: Testing Automated Echocardiography
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Principal Investigator, Emily MacKay, DO, MSHP, Assistant Professor, University of Pennsylvania
Other Study IDs: 848896
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: This Study is Being Conducted to Collect Echocardiographic Data to Test the Lumify Ultrasound With Hemodynamic Automation Device
Keywords: Philips Ultrasound; Ultrasound; Lumify Ultrasound; Hemodynamic Automation device; Lumify Ultrasound with Hemodynamic Automation; Automated hemodynamic output; Point-of-care echocardiographic imaging; Cardiac Surgery; Aortic valve repair; Mitral valve repair; Aortic valve replacement; Mitral valve replacement; Tricuspid valve repair; Tricuspid valve replacement; Pulmonic valve repair; Pulmonic valve replacement; Ascending aorta replacement; Coronary Artery Bypass Graft; Imaging
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Patient undergoing a cardiac surgery: Patients undergoing cardiac surgeries listed in inclusion criteria will be in this group.
  Interventions: Diagnostic Test: Ultrasound imaging
- Clinicians: Clinicians defined as physicians (e.g. attendings, fellows, residents) or advanced practice providers (e.g. nurse practitioners and physician assistants) will be in this group.

INTERVENTIONS:
Diagnostic Test: Ultrasound imaging — The intervention is non-invasive, chest wall, echocardiographic image acquisition in the cardiac operating room prior to a scheduled cardiac surgery. Echocardiographic images will be taken at three, key, timepoints in the operating room prior to cardiac surgery:
  1. Pre-induction.
  2. Post-induction / Pre-PAC
  3. Post-induction / Post-PAC
  Other Names: Philips Ultrasound; Lumify Ultrasound; Hemodynamic Automation device
  Groups: Patient undergoing a cardiac surgery

SUMMARY:
The purpose of this research is to determine if software can accurately predict certain heart parameters from chest wall ultrasound (non-radiation, non-invasive, imaging modality). An approved ultrasound device (Lumify) will be used to obtain images prior to cardiac surgery.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single visit clinical study. No additional interventions or follow-ups to the subject will be conducted as part of the study. All investigational scanning will be conducted using the as low as reasonably achievable (ALARA) principle to ensure the safety of the subjects. As ultrasound imaging is based on non-ionizing radiation, it is generally considered safe when used by appropriately trained health care providers. The study population will be adults. There are no specific enrollment targets, however it is expected that 120 subjects or fewer will be scanned to obtain the required 40 echocardiographic exams to complete this study. Exceeding the enrollment target of 120 subjects will require an amendment to the protocol. It is estimated this study will last for 12 months, at that time it will be evaluated and may potentially be amended.

This study is considered non-significant risk. There is no specific benefit to individuals participating in the study, however the feedback received is used to improve Philips systems and that can lead to increased diagnostic ability in future products.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and capable of providing informed consent and physically capable of performing study related activities
* Patient undergoing any of the following types of cardiac surgeries:

Aortic valve repair Aortic valve replacement Mitral valve repair Mitral valve replacement Tricuspid valve repair Tricuspid valve replacement Pulmonic valve repair Pulmonic valve replacement Ascending aorta replacement Coronary Artery Bypass Graft (CABG) surgery

Exclusion Criteria:

* Pregnant women
* Patients known to be under the jurisdiction of the Department of Corrections
* Patients with persistent arrhythmias as confirmed by the principal investigator (MacKay) on a caseby-case basis (e.g. atrial fibrillation, atrial flutter, frequent premature ventricular contractions, frequent premature atrial contractions, etc.)
* Patients with a contraindication to Pulmonary Arterial Catheter (PAC) monitoring as confirmed by the principal investigator (MacKay) on a case-by-case basis (e.g. tricuspid or pulmonic valve endocarditis, venous thrombosis present in the superior vena cava, right atrium, or main pulmonary artery)
* Patients with a contraindication to TEE monitoring as confirmed by the principal investigator (MacKay) on a case-by-case basis (e.g. previous esophageal surgery, prior gastric bypass surgery, esophageal varices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing predefined cardiac surgeries
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Correlation Testing Lumify Ultrasound with Hemodynamic Automation | 08/01/2021 - 08/31/2022
  Correlation between the hemodynamic parameters (e.g. stroke volume, cardiac output, cardiac index) obtained from the Lumify Ultrasound with Hemodynamic Automation with same hemodynamic parameters obtained from the reference standard of transesophageal echocardiography and pulmonary arterial catheterization by a single echocardiographer.
Repeatability (intraobserver variability) of hemodynamic parameters obtained from the Lumify Ultrasound with Hemodynamic Automation | 08/01/2021 - 08/31/2022
  Repeatability of the hemodynamic parameters (e.g. stroke volume, cardiac output, cardiac index) obtained from the Lumify Ultrasound with Hemodynamic Automation at set time intervals of one minute by a single echocardiographer.
Reproducibility (interobserver variability) of hemodynamic parameters obtained from the Lumify Ultrasound with Hemodynamic Automation | 08/01/2021 - 08/31/2022
  Reproducibility of the hemodynamic parameters (e.g. stroke volume, cardiac output, cardiac index) obtained from the Lumify Ultrasound with Hemodynamic Automation at set time intervals of one minute by a multiple echocardiographers blinded to each other's data.

SECONDARY OUTCOMES:
Clinical Efficacy of hemodynamic parameters obtained from the Lumify Ultrasound with Hemodynamic Automation | 08/01/2022 - 08/31/2023
  Clinician providers will evaluate the clinical efficacy of hemodynamic parameters obtained from the Lumify Ultrasound with Hemodynamic Automation by survey questions directly comparing the Lumify echocardiographic imaging to the reference standard

CONTACTS AND LOCATIONS:
Overall Officials: Roderic G Eckenhoff, MD, Study Chair — University of Pennsylvania, Department of Anesthesiology and Critical Care
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided